CLINICAL TRIAL: NCT05913531
Title: Retrospective Evaluation of Delirium Data From Previous Study Patients for Studies at the Clinic for Anesthesiology and Intensive Care Medicine CCM/CVK/CBF
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Intensive Care Medicine CCM/CVK/CBF, Charité - University Berlin, Charite University, Berlin, Germany
Other Study IDs: Retro-Delirium
Record Dates: First submitted 2023-05-11; First posted 2023-06-22 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of several studies of the Clinic for Anesthesiology and Intensive Care Medicine CCM/CVK/CBF to create a register with the delirium data from anesthesiology study patients between 18 - 100 years. The primary purpose of the register is to assess factors influencing the development of delirium.

In a subproject, risk factors that may lead to the development of postoperative delirium in the elderly will be evaluated with regard to gender differences using patients from the age of 60 with different surgical procedures. The risk factors examined are based on the evidence-based and consensus-based recommendations of the ESA guideline and literature review. In addition, the delirium incidence rate and the delirium severity is examined regarding gender differences.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age ≥ 18 years of studies of the clinic for Anesthesiology and Intensive Care Medicine CCM/CVK/CBF

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical male and female patients age ≥ 18 years of studies of the clinic for Anesthesiology and Intensive Care Medicine CCM/CVK/CBF
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Delirium | Up to 5 years
  Validated delirium scoring (points, duration and severity)

SECONDARY OUTCOMES:
Sedation scales | Up to 5 years
  Sedation is measured by the Richmond Agitation Sedation Scale
Socioeconomic information 1 | Up to 5 years
  Soci-economic information is collected by FIMA
Socioeconomic information 2 | Up to 5 years
  Soci-economic information is collected by the Nikolaus-score (social situation), 1. Subscale
Socioeconomic information 3 | Up to 5 years
  Soci-economic information is collected by items on socioeconomic status from the Federal Health Survey of 1998
Comorbidities | Up to 5 years
  Comorbidities are new diagnoses from hospital records.
Charlson comorbidity index | Up to 5 years
  Comorbidity scores
Lifestyle risks 1 | Up to 5 years
  Consumption of alcohol is measured by AUDIT (Alcohol Use Disorders Identification Tests)
Lifestyle risks 2 | Up to 5 years
  Consumption of and nicotine is measured by Fagerström Test for Cigarette Dependence (FTCD). Questionnaire scored 0-10 points with Total Score equal to the sum of all points
Lifestyle risks 3 | Up to 5 years
  Consumption of nicotine is measured by Smocking Pack Years (SPY)
Lifestyle risks 4 | Up to 5 years
  Previous consumption of nicotine is measured by History of Smoking.
Level of education | Up to 5 years
  Level of education is measured by ISCED (International Standard Classification of Education)
Quality of life - relatives | Up to 5 years
  Quality of life is measured by CarerQoL
Quality of life - self 1 | Up to 5 years
  Quality of life is measured by EQ-5D.An index calculated from the five EQ-5D (3L and 5L) dimensions by attaching specific weights to each severity level in each dimension.
Quality of life - self 2 | Up to 5 years
  Quality of life is measured by WHO-5. WHO-5 is a short and generic global rating scale measuring subjective well-being, the respondent is asked to rate how well each of the 5 statements applies to him or her when considering the last 14 days. Each of the 5 items is scored from 5 (all of the time) to 0 (none of the time). The raw score ranges from 0 (absence of well-being) to 25 (maximal well-being). Scores are then converted to a percentage scale from 0 (absent) to 100 (maximal). Higher scores represent greater psychological well-being.
Quality of life - self 3 | Up to 5 years
  Quality of life is measured by SF-12 (Short form health survey)
Functional impairment (IADL) 1 | Up to 5 years
  Instrumental Activities of Daily Living (IADLs) < 8
Functional impairment (ADL) 2 | Up to 5 years
  Activities of Daily Living (ADLs) < 100
Depression 1 | Up to 5 years
  Depression 1 is measured by PHQ-8 (Patient Health Questionnaire depression scale)
Depression 2 | Up to 5 years
  Depression 2 is measured by GDS (Geriatric Depression Scale)
Depression 3 | Up to 5 years
  Depression 3 is measured by HADS (Hospital Anxiety and Depression Scale)
Depression 4 | Up to 5 years
  Depression 4 is measured by CDS (Cornel Depression Scale)
Anxiety scales 1 | Up to 5 years
  Anxiety is measured by GAD-7 (Generalized Anxiety Disorder 7)
Anxiety scale 2 | Up to 5 years
  Anxiety 2 is measured by FAS (Faces Anxiety Scale)
Anxiety scale 2 | Up to 5 years
  Anxiety 2 is measured by GAD-7
Pain | Up to 5 years
  Pain is measured by numeric pain scales (minimum = 0, maximum = 10).
Type of concomitant medication | Up to 5 years
  The medication administered during the hospital stay is documented.
Anticholinergic Load | Up to 5 years
  Measured by anticholinergic drug scale
Frailty | Up to 5 years
  Frailty is measured with a modified frailty score according to Fried´s frailty phenotype assessment.
Nutritional status 1 | Up to 5 years
  Nutritional status 1 is measured by calf circumference
Nutritional status 2 | Up to 5 years
  Nutritional status 2 is measured by arm circumference
Nutritional status 3 | Up to 5 years
  Nutritional status 3 is measured by changes in weight
Nutritional status 4 | Up to 5 years
  Nutritional status 4 is measured by changes in body mass index
Nutritional status 5 | Up to 5 years
  Nutritional status 5 is measured by previous weight history (3 months)
Nutritional status 6 | Up to 5 years
  Nutritional status 6 is measured by Medi-Score
Nutritional status 7 | Up to 5 years
  Nutritional status 7 is measured by MNA-SF
Nutritional status 8 | Up to 5 years
  Nutritional status 8 is measured by Sarcopenia
Nutritional status 9 | Up to 5 years
  Nutritional status 9 is measured by Nutritional Risk Screening (NRS 2002)
Nutritional status 10 | Up to 5 years
  Nutritional status 10 is measured by AKE Screening
Mobility 1 | Up to 5 years
  Mobility 1 is measured with the Timed up and Go
Mobility 2 | Up to 5 years
  Mobility 2 is measured with a walking test: Slowness: Calculated after walking 3 meters, adjusted for sex and height, according to Fried. The cut-off points for 3 meters were established as, in men: height ≤173 cm and time ≥4.59 s (equivalent to 0.65 m/s); height >1.73 cm and time ≥3.93 s (equivalent to 0.76 m/s); and for women: height ≤1.59 cm and time ≥4.59 s (0.65 m/s); and height >1.59 cm and time ≥3.93 s (0.76 m/s).
Number of participants with changes in laboratory values 1 | Up to 5 years
  Laboratory results in the hospital including hemoglobin, lymphocytes, total neutrophils, platelet count, white blood cell (WBC) count and inflammatory markers from blood samples.
Number of participants with changes in laboratory values 2 | Up to 5 years
  Laboratory results in the hospital from serum samples
Number of participants with changes in laboratory values 3 | Up to 5 years
  Laboratory results in the hospital from urine samples
Number of participants with changes in laboratory values 4 | Up to 5 years
  Laboratory results in the hospital from liquor samples
Depth of sedation | Up to 5 years
  The sedation was measured intraoperatively processed electroencephalogram (EEG) Full-brain EEG recording with surface electrodes, raw EEG analysis measured during the operation.
Type of operation | Up to 5 years
  Type of operation is measured by OPS-Code
Duration of operation | Up to 5 years
  Type of operation is measured in minutes
Type of anesthesia | Up to 5 years
  There are four main categories of anesthesia used during surgery and other procedures: general anesthesia, regional anesthesia, sedation (sometimes called "monitored anesthesia care"), and local anesthesia.
Duration of anesthesia | Up to 5 years
  Duration of anesthesia is measured in minutes.
Length of hospital stay | Up to 5 years
  Hospital stay is measured in days.
Intensive care unit stay | Up to 5 years
  Intensive care unit stay is measured in hours.
Organ complications | Up to 5 years
  Organ complications are recorded in hospital records
Hospital discharge criteria | Up to 5 years
  Discharge criteria are measured at hospital discharge by Post Anesthetic Discharge Scoring System (PADS) Score
Mortality | Up to 5 years
  Mortality rate is measured after 1,2,3,4 and 5 years
Study data | Up to 5 years
  Identification of study data with a high impact on delirium from the study databases
Sleeping items | Up to 5 years
  Questions measuring personal satisfaction with sleep quality and duration As measured by questions measuring personal satisfaction with sleep quality and duration
Circadian rhythm variables | Up to 5 years
  Items measuring circadian rhythm variables e.g. Zeitgebers

OTHER OUTCOMES:
Parameter of cognition | Up to 5 years
  Cognitive functioning will be measured with a battery of computerized neuropsychological tests.
Parameter of cognition | Up to 5 years
  Cognitive functioning will be measured with a battery of non-computerized neuropsychological tests.
Demographic data | Up to 5 years
  Demographic data are documented in the hospital records.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anaesthesiolgy and Intensive Care Medicine CVK/CCM, Charité - Univeristy Medicine Berlin, Berlin, Germany